CLINICAL TRIAL: NCT05585762
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Feasibility Pilot Study to Evaluate the Tolerability and Safety of a Novel Ketone Ester Ingredient in Healthy Older Men and Women.
Brief Title: Buck Institute Ketone Ester RCT
Acronym: BIKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buck Institute for Research on Aging (Other)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BUCK_2201
Record Dates: First submitted 2022-10-03; First posted 2022-10-19 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-01

CONDITIONS: Tolerance; Safety Issues; Aging
Keywords: Ketone ester; Tolerance; Safety; Aging
MeSH Terms: interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Parallel group, randomized, double-blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study products will be allocated a code and labelled by an external team. The coding of the study products will be recorded and sealed in 'unblinding envelopes' that will only be opened in unblinding becomes necessary for subject safety. No one on the study team (including outcome assessor and statisticians) will be aware of the study product identity. The study products are matched for appearance, taste and calories and will not be visibly distinguishable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone ester (Experimental): Flavored ketone ester beverage 75 mL. Day 0 - 7: half of one bottle consumed daily. Day 8 to end (Week 12): one full bottle consumed daily.
  Interventions: Other: Ketone ester
- Non-ketone placebo (Placebo Comparator): Flavored beverage with bitter additive 75 mL. Matched for appearance, taste and calories. Day 0 - 7: half of one bottle consumed daily. Day 8 to end (Week 12): one full bottle consumed daily.
  Interventions: Other: Non-ketone placebo

INTERVENTIONS:
Other: Ketone ester — 75 mL chocolate flavored beverage containing 25 g of ketone ester. Half a bottle (12.5 g/day) will be consumed for the first 7 days and a complete bottle (25 g/day) will be consumed for the remaining 77 days.
  Arms: Ketone ester
Other: Non-ketone placebo — 75 mL chocolate flavored beverage containing 25 g of non-ketogenic fat. Half a bottle (12.5 g/day) will be consumed for the first 7 days and a complete bottle (25 g/day) will be consumed for the remaining 77 days.
  Arms: Non-ketone placebo

SUMMARY:
This study is to investigate the tolerability and safety of a ketone promoting ingredient, called a ketone ester (KE), in healthy older adults. This randomized, double-blind, placebo-controlled trial aims to characterize the tolerability and safety of daily consumption of the KE in healthy older adults (over 65 years old) over 12 weeks. Study participants will complete Beverage Tolerability Questionaires (BTQ) to rate any side side effects throughout the study. Safety will also be assessed by collection of blood and urine samples, vital signs, body weight, and monitoring of adverse events (AEs). The study will also collect pilot data to explore possible effects of KE on physical function, cognitive function and quality of life. The findings of this study will be used to facilitate future mechanistic studies of KE in aging.

DETAILED DESCRIPTION:
Screening (Phone and Visit 1): Subjects are screened for eligibility by telephone for major exclusion criteria. They then attend a screening visit. At the start of the visit subjects must meet pre-test requirements (fasting ≥ 10 h, no alcohol ≥ 10 h, no exercise ≥ 10 h, no cannabis products ≥ 10 h). During this visit, consent is obtained, followed by a medical history interview, a physical assessment (including vital signs, body weight, and waist circumference) and fasting blood samples are collected for screening analysis of: clinical chemistry, hematology, lipid profile, thyroid hormones. A clean catch urine sample is also collected for urinalysis. Subjects eligible and willing to take part in the study are randomized to take one of the two ketone ester serving sizes (12.5 g , 25 g) for the ketone kinetics visit (Visit 2). Subjects will be given a stool sample collection kit to take home for at-home sample collection up to 3 days before Visit 2, the stool sample will be returned to investigators using a prepaid mailer.

Ketone Kinetics Visit (Visit 2): Subjects must meet pre-test requirements (as above). A BTQ (Beverage Tolerability Questionnaire) is used to observe the tolerability of ketone drinks before and after their consumption. Blood glucose and ketone levels are measured from a finger stick sample of a ketone meter at baseline, and at 30, 60, 90,120,180, 240-minute timepoints. Subjects are then randomized to their experimental group ketone ester or placebo for the remainder of the visits (Visit 3-5). Subjects will be given a stool sample collection kit to take home for at-home sample collection up to 3 days before Visit 3; samples are returned by mail.

Baseline Visit (Visit 3- Week 0): Subjects must meet pre-test requirements (as above). Fasted blood samples are collected for screening analysis of: clinical chemistry, hematology, lipid profile, thyroid hormones. A clean catch urine sample is collected for screening analysis and urinalysis and additional plasma is banked for future aging biomarker analysis. Subjects will undergo an interview for Katz's Activities of Daily Living (ADL), and Lawton's Instrumental Activities of Daily Living (IADLs), and CSHA Frailty Score (Canadian Study of Health and Aging). Subjects also complete the following paper questionnaires: Profile of Mood States (Short form), The Sexual Quality of Life Questionnaire (Male or Female Version), Short Form Health Survey-36, Pittsburgh Sleep Quality Index, Pittsburgh Fatiguability Scale and Geriatric Depression Scale. Physical and cognitive measures are assessed through the following tests: Montreal Cognitive Assessment, Digit Symbol Substitution Task and Trails A and B. Subjects also complete physical function testing at baseline (Visit 3) and final visit (Visit 5): Short Physical Performance Battery, 1 rep max leg press, sub maximal leg press repetitions to failure, 6-minute walk test and grip strength.

At the end of the testing, a continuous glucose and ketone monitor is applied (lasting 2 weeks). Subjects will be given a stool sample collection kit to take home for at-home sample between Week 1 and 2; samples are returned by mail. Subject will be given a month's supply of study product to take home. Subjects will be reminded of study instructions (for study beverage consumption, daily Study Log completion, and to maintain habitual exercise, meal/diet, and medication/supplementation use).

At home procedures (Week 0 - 12): Each day at home, subjects should consume their first meal of the day at a similar time and consume the study product within 5 minutes of finishing their first meal. Subjects will complete the Study Log immediately before they consume their second meal of the day or a snack (3 - 6 h after the study beverage). For Days 1 - 14 the Study Log will query the presence of specific symptoms with a beverage tolerance questionnaire (BTQ) and will confirm that subjects consumed their study product. From Day 15 onwards, the Study Log records study product consumption, but a full BTQ is not completed; however, any symptoms can be noted to assess tolerance by interview for the previous 2-week interval; at Visit 4- Week 4, during phone check-ins (Week 5, 8, and 10) and at Visit 5. At Week 8, subjects will be mailed the final mont's supply of study product, a continuous glucose and ketone sensor to apply at home (Week 10), and a stool sample collection kit for at-home sample collection up to 3 days before Visit 5 (Week 12), samples are returned by mail.

Intermediate Visit (Visit 4- Week 4): Subjects must meet pre-test requirements (as above). Fasted blood samples are collected for screening analysis of: clinical chemistry, hematology, lipid profile, thyroid hormones. A clean catch urine sample is collected for screening analysis and urinalysis and additional plasma is banked for future aging biomarker analysis. Tolerance of the study beverage and Adverse Events are assessed by interview. Subjects will be given a month's supply of study product to take home. Subjects will be given a stool sample collection kit to take home for at-home sample collection up to 3 days after Visit 4; samples are returned by mail.

Final Visit (Visit 5- Week 12): Follows identical testing procedures to Baseline Visit (Visit 3, Week 0).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 65 years of age, inclusive at Visit 1.
2. Subject has a BMI 18.5-34.9 kg/m2 (inclusive) at Visit 1.
3. Subject is willing and able to comply with all study procedures including randomization into any of the experimental groups, maintenance of habitual dietary intake, exercise and medication and supplement use, blood draws and the following prior to test visits: fasting (≥10 h; water and black coffee only), no alcohol (≥ 10 h), no cannabis products (≥10 h) and no exercise (≥ 10 h).
4. Subject has no health conditions that would prevent them from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
5. Subject understands the study procedures and signs forms providing informed consent to participate in the study.

Exclusion Criteria:

1. Subject is non ambulatory
2. Subject has a CSHA clinical frailty score > 5
3. Subject requires assistance with any activity of daily living
4. Subject lives in an institutional setting (skilled nursing facility or residential care facility for the elderly).
5. Subject is a female who has not passed menopause.
6. Subject is unable to converse in English
7. Subject is unable to provide informed consent due to cognitive impairment or insufficient English language comprehension
8. Subject has been hospitalized within 30 days of Visit 1, 2 or 3.
9. Subject has an abnormal laboratory test result(s) of clinical importance, indicating unstable chronic disease of major organ dysfunction, at Visit 1, at the discretion of the Medical Officer. One re-test will be allowed on a separate day prior to Visit 2, for subjects with abnormal laboratory test results.
10. Subject has a history or presence of uncontrolled and/or clinically active pulmonary, cardiac (e.g. >= New York Heart Association class III), hepatic, renal, endocrine (including type 1 diabetes), hematologic, immunologic, neurologic (e.g., Alzheimer's or Parkinson's diseases), psychiatric (including unstable depression and/or anxiety disorders) or biliary disorders. Stable chronic disease is not an exclusion criterion unless specified.
11. Subject has a clinically important gastrointestinal condition that would potentially interfere with the evaluation of the study beverage [e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation, severe constipation (in the opinion of the Clinical Investigator), history of frequent diarrhea, history of surgery for weight loss, gastroparesis, systemic disease that might affect gut motility according to the Investigator, reflux requiring daily medication, history of gastrointestinal ulcers or bleeding, and/or clinically important lactose intolerance].
12. Subject has a history of alcohol or substance abuse.
13. Subject is consistently using prescriptive or over-the counter medications where alcohol is a contraindication at the discretion of the Investigator.
14. Subject has a known allergy, intolerance, or sensitivity to any of the ingredients in the study beverages, including soy and milk protein.
15. Subject has uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1. One re-test will be allowed on a separate day before Visit 2, for subjects with abnormal blood pressure.
16. Subject is undergoing treatment or active surveillance for cancer, or has been diagnosed with cancer in the prior two years, except for non-melanoma skin cancer.
17. Subject has recently used antibiotics within 30 days of Visit 1, 2 or 3.
18. Subject has extreme dietary habits (e.g., intermittent fasting or time restricted eating, Atkins diet, vegan, very high protein/low carbohydrate or has used weight-loss medications (including over-the-counter medications and/or supplements) or programs within 30 days of Visit 1, 2 or 3.
19. Subject has used medications (over-the-counter or prescription) known to influence gastrointestinal function including, but not limited to, opioids, weight loss medications, antidiarrheals, and antispasmodics) within 30 days of Visit 1, 2 or 3.
20. Subject has used ketone supplements (ketone salts or esters, and medium chain triglycerides [MCT]) within 30 days of Visit 1, 2 or 3.
21. Subject has unstable use of thyroid, antihypertensive, antidepressant, or statin medications within 30 days of Visit 1, 2 or 3.
22. Subject has a condition the Clinical Investigator believes would interfere with their ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.
23. Subject works nights or shifts that means it is not possible to maintain a consistent meal schedule during the study.
24. Subject is not permitted to visit the Buck Institute campus, for example due to inability to confirm COVID-19 vaccination status.
25. Subject does not have a Bluetooth enabled smartphone.
26. Subject does not have access to the internet

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Tolerance | 12 weeks
  The primary outcome measure is the proportion of subjects reporting the same moderate to severe symptom (among dizziness, headache or nausea) occurring on more than one day within any given recall period (after week 0 - 2 acclimation period) when ketone esters are consumed daily for 12 weeks.

SECONDARY OUTCOMES:
Safety Blood Profile | Change from baseline to week 4, and week 12.
  Change from baseline to week 4 and week 12 in the incidence of abnormal laboratory test results
Ketone changes 4h after ketone ester drinks | 4 hours
  Subjects consume a single serving of either 12.5 g or 25 g of ketone ester. After this, their short-term (regularly over 4h) blood ketone changes are measured using capillary blood sampling.

OTHER OUTCOMES:
Change in Short Physical Performance Battery Score | Measured at baseline (Week 0) and final visit (Week 12)
  Standard set of tests to measure physical function in elderly
Change in 1 rep max leg press | Measured at baseline (Week 0) and final visit (Week 12)
  Heaviest weight moved using leg press machine
Change in Sub maximal leg press to fatigue | Measured at baseline (Week 0) and final visit (Week 12)
  Number of reps completed at a sub maximal weight
Change in 6 minute walk test | Measured at baseline (Week 0) and final visit (Week 12)
  Distance covered when walking for 6 minutes
Change in Grip strength | Measured at baseline (Week 0) and final visit (Week 12)
  Hand grip force measured by dynamometer
Change in Montreal Cognitive Assessment score | Measured at baseline (Week 0) and final visit (Week 12)
  Standard test for cognitive function in elderly
Change in Digit Symbol Substitution Task scores | Measured at baseline (Week 0) and final visit (Week 12)
  Task where participant substitutes numbers for symbols in a set time
Change in Trails A and B scores | Measured at baseline (Week 0) and final visit (Week 12)
  Standard trail making test scores between letters and numbers
Change in score on Profile of Mood States (Short form) Questionnaire | Measured at baseline (Week 0) and final visit (Week 12)
  Questionnaire
Change in score on The Sexual Quality of Life Questionnaire | Measured at baseline (Week 0) and final visit (Week 12)
  Questionnaire
Change in score on the Short Form Health Survey-36 | Measured at baseline (Week 0) and final visit (Week 12)
  Questionnaire
Change in score on the Pittsburgh Sleep Quality Index | Measured at baseline (Week 0) and final visit (Week 12)
  Questionnaire.
Change in score on the Pittsburgh Fatiguability Scale | Measured at baseline (Week 0) and final visit (Week 12)
  Questionnaire
Change in score on the Geriatric Depression Scale | Measured at baseline (Week 0) and final visit (Week 12)
  Questionnaire
Changes in gut microbial diversity | Change from pre-test to week 1, week 4 and week 12.
  DNA sequencing of bacterial species in stool samples.
Ketone changes 4h after powder formulation of ketone drinks | 4h
  Subjects consume a single serving of either 12.5 g or 25 g of powder formulation ketone ester. After this, their short-term (regularly over 4h) blood ketone changes are measured using capillary blood sampling.

CONTACTS AND LOCATIONS:
Overall Officials: John C Newman, MD, PhD, Principal Investigator — Buck Institute
Locations (1):
- Buck Institute for Research on Aging, Novato, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen O, Blonquist TM, Mah E, Sanoshy K, Beckman D, Nieman KM, Winters BL, Anthony JC, Verdin E, Newman JC, Stubbs BJ. Tolerability and Safety of a Novel Ketogenic Ester, Bis-Hexanoyl (R)-1,3-Butanediol: A Randomized Controlled Trial in Healthy Adults. Nutrients. 2021 Jun 16;13(6):2066. doi: 10.3390/nu13062066. PMID 34208742
- [Background] Crabtree CD, Blade T, Hyde PN, Buga A, Kackley ML, Sapper TN, Panda O, Roa-Diaz S, Anthony JC, Newman JC, Volek JS, Stubbs BJ. Bis Hexanoyl (R)-1,3-Butanediol, a Novel Ketogenic Ester, Acutely Increases Circulating r- and s-ss-Hydroxybutyrate Concentrations in Healthy Adults. J Am Nutr Assoc. 2023 Feb;42(2):169-177. doi: 10.1080/07315724.2021.2015476. Epub 2022 Mar 25. PMID 35512774
- [Derived] Stubbs BJ, Stephens EB, Mansfield T, Senadheera C, Diaz SR, Peralta S, Alexander L, Silverman-Martin W, Kurtzig J, Fernando BA, Garcia TY, Yukawa M, Morris J, Yurkovich JT, Newman AB, Johnson JB, Cawthon PM, Newman JC. Exploratory functional and quality of life outcomes with daily consumption of the ketone ester bis-octanoyl (R)-1,3-butanediol in healthy older adults: a randomized, parallel arm, double-blind, placebo-controlled study. J Frailty Aging. 2025 Dec;14(6):100106. doi: 10.1016/j.tjfa.2025.100106. Epub 2025 Nov 27. PMID 41313689
- [Derived] Stubbs BJ, Stephens EB, Senadheera C, Diaz SR, Peralta S, Alexander L, Silverman-Martin W, Kurtzig J, Fernando BA, Yurkovich JT, Garcia TY, Yukawa M, Morris J, Johnson JB, Newman JC. Exploratory functional and quality of life outcomes with daily consumption of the ketone ester bis-octanoyl (R)-1,3-butanediol in healthy older adults: a randomized, parallel arm, double-blind, placebo-controlled study. medRxiv [Preprint]. 2024 Sep 18:2024.09.17.24313811. doi: 10.1101/2024.09.17.24313811. PMID 39371165
- [Derived] Stubbs BJ, Stephens EB, Senadheera C, Peralta S, Roa-Diaz S, Alexander L, Silverman-Martin W, Garcia TY, Yukawa M, Morris J, Blonquist TM, Johnson JB, Newman JC. Daily consumption of ketone ester, bis-octanoyl (R)-1,3-butanediol, is safe and tolerable in healthy older adults in a randomized, parallel arm, double-blind, placebo-controlled, pilot study. J Nutr Health Aging. 2024 Sep;28(9):100329. doi: 10.1016/j.jnha.2024.100329. Epub 2024 Aug 12. PMID 39137624
- [Derived] Stubbs BJ, Stephens EB, Senadheera C, Peralta S, Roa-Diaz S, Alexander L, Silverman-Martin W, Garcia TY, Yukawa M, Morris J, Blonquist TM, Johnson JB, Newman JC. Daily consumption of ketone ester, bis-octanoyl (R)-1,3-butanediol, is safe and tolerable in healthy older adults, a randomized, parallel arm, double-blind, placebo-controlled, pilot study. medRxiv [Preprint]. 2024 May 5:2024.05.03.24306699. doi: 10.1101/2024.05.03.24306699. PMID 38746215